CLINICAL TRIAL: NCT05883826
Title: The Effect of Sexual Health Training Given to Nursing Students With the PLISSIT Model on Knowledge and Attitude
Brief Title: The Effect of Sexual Health Training Given to Nursing Students on Knowledge and Attitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, CEYDA SU GUNDUZ, Study director, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: marmaraceydasugunduzistanbul34
Record Dates: First submitted 2023-04-07; First posted 2023-06-01 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Nursing Education; Nursing Students; Nursing Model

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLISSIT Group (Experimental): Nursing students in this group will be given sexual health training. The training will last for 4 weeks. The training is 16 hours in total. During the training, students will learn the PLISSIT model and evaluate cases involving using this model. Questionnaire will be applied before the training, immediately after the training and 3 months after the training.
  Interventions: Behavioral: sexual health training
- Control group (No Intervention): Nursing students in this group will not be subjected to any application and will continue their routine nursing lessons. The questionnaire will be administered to the control group before the training given to the experimental group, immediately after the training and 3 months after the training.

INTERVENTIONS:
Behavioral: sexual health training — The 16-hour sexual health training will be given for 4 weeks. Case discussions using the PLISSIT Model will be held in the training content.
  Arms: PLISSIT Group

SUMMARY:
Nurses play an important role in providing sexual health care to individuals. In this study, sexual health education will be implemented in an innovative way by supporting the use of models in the process of sexual counseling of nursing students to patients. The PLISSIT model, which is most frequently used when providing sexual counseling services to patients, will be taught to nursing students and its effectiveness will be determined. In the literature, only one study was found regarding the use of the PLISSIT model in sexual health assessment, conducted with students. The research was planned as pretest-posttest comparative, randomised, with an experimental and a control group, and with repeated measurements, in order to determine the effect of sexual health education given to nursing students with the PLISSIT model on sexual health care knowledge, sexual health care attitudes and myths about sexual health. This research will be carried out between December 2023 and March 2024 with the participation of fourth-year students studying at Marmara University, Faculty of Health Sciences, Department of Nursing. Students who meet the inclusion criteria will be randomly assigned to experimental (n=45) and control (n=45) groups. The data of the research will be obtained using the "Student Information Form", "Knowledge of Sexual Healthcare Scale ", "Attitude to Sexual Healthcare Scale", "Sexual Myths Scale" and "Student Opinion Form on Sexual Health Education". Ethical permission and institutional permission were obtained. The research While routine training will be given to the control group during the training, the experimental group will be given sexual health training including 16 hours of PLISSIT model teaching by the researcher. The data of the research will be obtained before the training, immediately after the training and 3 months after the training, using a data collection form.

DETAILED DESCRIPTION:
Sexuality is a central aspect of being human that encompasses all life. Nurses play an important role in providing sexual health care to individuals. There is evidence in the literature that the knowledge and skills that nurses should have in order to provide sexual health care are not sufficient. The main reason why nurses have problems in the provide sexual health care is that the subject of sexuality is not sufficiently included in the undergraduate nursing education. Sexual health education programs should be structured in a way to effectively increase the competencies of nursing students. The use of models in sexual counseling enables students to relate theory and practice to sexual health care. In this study, sexual health training will be implemented in an innovative way by supporting the use of models in the process of providing sexual counseling to the patients of nursing students. The most commonly used PLISSIT model will be taught to nursing students while providing sexual counseling to patients and its effectiveness will be determined. In the literature, only one study was found with students on the use of the PLISSIT model in sexual health assessment. The research is planned to be pre-test post-test comparative, randomized, with one experiment and one control group, repeated measurement ın order to determine the effect of the sexual health training given to nursing students with the PLISSIT model on the myths about sexuality, sexual health care knowledge and sexual health care attitude. This research will be carried out between December 2023 and March 2024 with the participation of fourth grade students studying at Marmara University Faculty of Health Sciences, Department of Nursing. Students who is suitable the inclusion criteria will be randomized to the experimental (n=45) and control groups (n=45). The data of the research will be obtained by using "Student Information Form", "Sexual Health Care Knowledge Scale", "Sexual Health Care Attitude Scale" and "Sexual Myths Scale" and "Student Opinion Form on Sexual Health Education". Ethical permission and institutional permission were obtained.During the research, while the control group receives routine training, the experimental group will be given a sexual health assessment training including 16 hours of PLISSIT model teaching by the researcher. The data of the research will be obtained by using the data collection form before the training, immediately after the training and 3 months after the training. By ensuring that nursing students learn and practice sexual health assessment, the sexual health of individuals will be protected and improved.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior nursing student,
* Having sufficient Turkish speaking and understanding skills,
* Agreeing to participate in sexuality education on the online platform if necessary,
* Sufficient or unlimited internet access,
* Having any computer, tablet or smart phone,
* Being willing to participate in the research

Exclusion Criteria:

* Desire to leave the research,
* Incomplete filling of data collection forms,
* Not attending more than 30% of the training given in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Sexual Healthcare Scale | baseline
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "I don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Knowledge of Sexual Healthcare Scale | week 4
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "I don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Knowledge of Sexual Healthcare Scale | month 3
  The scale was designed to measure the knowledge of nursing students about sexual health care. The scale consists of 31 items. Each item was rated as "yes", "no" and "I don't know". 1 point is given for the correct answer, 0 points for the wrong answer and the answer I don't know. A score between 0-31 can be obtained from the scale.
Attitude to Sexual Healthcare Scale | baseline
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 sub-dimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.
Attitude to Sexual Healthcare Scale | week 4
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 sub-dimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.
Attitude to Sexual Healthcare Scale | month 3
  The scale determines the attitudes of nursing students towards sexual health services. The scale consists of 3 sub-dimensions and a total of 18 questions. Each item on the 5-point Likert scale is rated as 5 = strongly agree, 4 = agree, 3 = undecided, 2 = disagree, and 1 = strongly disagree. The scores that can be obtained from the scale vary between 18 and 90.

SECONDARY OUTCOMES:
Sexual Myths Scale | baseline
  The scale has been reported to be a useful tool to reveal whether a person's knowledge is based on sexual myths. In this 5-point Likert-type scale, consisting of 28 items, statements are evaluated between "1" points (I never agree), "5" points (I totally agree). The scale consists of 8 sub-dimensions and 28 items. The total score that can be obtained from the scale can vary between 28-140.
Sexual Myths Scale | week 4
  The scale has been reported to be a useful tool to reveal whether a person's knowledge is based on sexual myths. In this 5-point Likert-type scale, consisting of 28 items, statements are evaluated between "1" points (I never agree), "5" points (I totally agree). The scale consists of 8 sub-dimensions and 28 items. The total score that can be obtained from the scale can vary between 28-140.
Sexual Myths Scale | month 3
  The scale has been reported to be a useful tool to reveal whether a person's knowledge is based on sexual myths. In this 5-point Likert-type scale, consisting of 28 items, statements are evaluated between "1" points (I never agree), "5" points (I totally agree). The scale consists of 8 sub-dimensions and 28 items. The total score that can be obtained from the scale can vary between 28-140.
Student Opinion Form on Sexual Health Education (part 1) | week 4
  It determines the thoughts of the students about the model taught in education and the satisfaction of the students from the education.
Student Opinion Form on Sexual Health Education (part 2) | month 3
  It determines the impact of education on providing sexual health care to individuals during intern internship of students.

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Demirci, Prof., Study Director — Marmara Üniversity
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No